CLINICAL TRIAL: NCT04672447
Title: Effects of 4 Weeks Supplementation With L-Citrulline and Glutathione on Arterial Function and Cardiovascular Responses in Postmenopausal Healthy Women: A Pilot Study
Brief Title: Effect of 4 Weeks of Citrulline and Glutathione Supplementation on Arterial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Kyowa Hakko Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-0152
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Menopause; Cardiovascular Risk Factor
Keywords: Endothelial Function; Aortic Hemodynamics; Pressure Wave Reflection
MeSH Terms: interventions — Citrulline; Glutathione

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment Masking: Double Blind (Subject, Investigator)
Who Masked: Participant, Investigator
Masking Description: Randomized, placebo-controlled, double-blind, parallel-groups study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-Citrulline + Glutathione (Experimental): Citrulline: 2 grams/day, Glutathione: 200mg/day for 4 weeks
  Interventions: Dietary Supplement: L-Citrulline; Dietary Supplement: Glutathione
- L-Citrulline (Experimental): Citrulline: 6 grams/day
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Maltodextrin: 6 grams/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — Four weeks of oral L-Citrulline (2 grams/day) supplementation. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: L-Citrulline + Glutathione
Dietary Supplement: L-Citrulline — Four weeks of oral L-Citrulline (6 grams/day) supplementation. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: L-Citrulline
Dietary Supplement: Placebo — Four weeks of oral placebo (6 grams/day maltodextrin) supplementation. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: Placebo
Dietary Supplement: Glutathione — Four weeks of Glutathione (200mg/day) supplementation. Supplementation will be ingested daily, half of the doses in the morning and half at night.
  Arms: L-Citrulline + Glutathione

SUMMARY:
Examining the effects of 4 weeks of Citrulline alone or in combination with glutathione on the arterial function of postmenopausal women.

DETAILED DESCRIPTION:
L-Citrulline is a non-protein amino acid and an efficient precursor of L-arginine, the substrate for endothelial nitric oxide synthesis. Glutathione is a tripeptide with antioxidant effects. Postmenopausal women will ingest 6g/d of L-Citrulline or 2g of L-Citrulline plus 200mg/d of glutathione or placebo (maltodextrin) for 4 weeks with vascular function testing prior to and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, postmenopausal women (defined as the absence of menstruation for at least 1 year).
2. Between the ages of 50-79 years.
3. Body mass index of 18.5 - 34.9 kg/m2.
4. Brachial systolic blood pressure < 150 mmHg, and diastolic blood pressure < 90 mmHg.
5. Sedentary (defined as < 120 min/week of exercise).
6. Be willing and able to comfortably abstain from any of food supplements for the period of time beginning 1 month prior to the study to the time of the termination of the study.
7. Not participating as a subject in another study for at least 2 months prior to the study and for the duration of this study.

Exclusion Criteria:

1. Current or prior use of tobacco products, e-cigarettes or other inhaled substance.
2. Use of medications and/or any supplements that may affect outcome variables (such as arginine-containing supplements, nitroglycerin, statin drugs, but not limited to those.)
3. Taking hormone replacement therapy during the 3 months before the study.
4. More than a moderate intake of alcohol (>7 drink per week).
5. Cardiovascular diseases, diabetes and other metabolic or chronic diseases.
6. Musculoskeletal disorders that will prevent exercise performance.
7. Currently taking more than one vasoactive drug for blood pressure control.

   * Subject having no more than one drug for prevention, which does not affect variables, may be included, but will be diagnosed as not having a disease.

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | 4 weeks
  Endothelial function will be measured before and after the intervention using brachial artery flow mediated dilation at rest, blood flow measured in the brachial artery during handgrip exercise, and blood flow in the common femoral artery during passive leg movement. All measurements performed using doppler ultrasound.
Change in arterial stiffness | 4 weeks
  Arterial stiffness will be assessed through measurement of pulse-wave velocity of the carotid-femoral, carotid radial, carotid-ankle and femoral ankle arterial segments before and after the 4 week interventions.
Blood pressure control during the cold pressor test | 4 weeks
  Blood pressure will be measured during the cold pressor test before and after the 4 weeks.
L-Arginine bioavailability | 4 weeks
  Plasma levels of arginine will be measured before and after the 4 week intervention.

SECONDARY OUTCOMES:
cardiovascular hemodynamics using pulse wave analysis during the cold pressor test | 4 weeks
  arterial tonometry will be measured during the cold pressor test before and after the 4 week intervention.
body composition | 4 weeks
  We will determine whether L-citrulline + glutathione changes body composition more than L-citrulline or placebo.
Muscle Strength | 4 weeks
  Leg Extension strength will be measured before and after the 4 weeks.
L-Citrulline levels | 4 weeks
  Plasma levels of L-Citrulline will be measured before and after the 4 weeks.
Glutathione peroxidase levels | 4 weeks
  Blood levels of glutathione peroxidase will be measured before and after the 4 weeks
Malondialdehyde | 4 weeks
  blood levels of malondialdehyde will be measured before and after the 4 weeks
L-Ornithine levels | 4 weeks
  plasma levels of L-ornithine will be measured before and after the 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- TTU Kinesiology and Sport Management Building, Lubbock, Texas, United States